CLINICAL TRIAL: NCT06062784
Title: Exploring the Utility of Bedside Tests for Predicting Cardiorespiratory Fitness in Older Adults
Brief Title: Bedside Tests of Cardiorespiratory Fitness
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: BedTestAge
Record Dates: First submitted 2023-09-07; First posted 2023-10-02 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Aging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A study of 64 older adults over the age of 65y to assess the utility of patient characteristics and bedside measures of physical function and muscle size to predict cardiorespiratory fitness.

DETAILED DESCRIPTION:
A study of 64 older adults over the age of 65y to assess the utility of patient characteristics (age, gender and BMI) and bedside measures of physical function (handgrip strength (HGS) and step box test) and muscle size (muscle thickness via B-mode ultrasonography (US)) to predict cardiorespiratory fitness (VO2peak and anaerobic threshold) as measured by the gold-standard assessment method, cardiopulmonary exercise testing (CPET).

Each participant will take part in a single assessment day (after health screening against CPET safety criteria) whereby they will have US measures of the vastus lateralis before completing HGS and step box test assessments, and finally a CPET.

ELIGIBILITY:
Inclusion Criteria:

* Over 65y
* Independent, community-dwelling

Exclusion Criteria:

* Contraindications to CPET safety criteria

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community dwelling adults over the age of 65y who were able to provide written, informed consent and had no contraindications to exercise testing.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory fitness (CRF) - VO2 max | Single time-point - 8 to 12 minutes
  CRF via cardiopulmonary exercise testing (CPET). This includes a measure of maximum oxygen uptake (VO2 max) determined via inline breath gas analysis during an incremental cycle test.
Cardiorespiratory fitness (CRF) - Anaerobic threshold | Single time-point - 8 to 12 minutes
  CRF via cardiopulmonary exercise testing (CPET). This includes a measure of anaerobic threshold (AT) determined via inline breath gas analysis during an incremental cycle test.

SECONDARY OUTCOMES:
Muscle architecture - muscle thickness | Single time-point: 10 minutes
  Analysis of vastus lateralis muscle thickness using b-mode ultrasonography
Muscle architecture - pennation angle | Single time-point: 10 minutes
  Analysis of vastus lateralis pennation angle using b-mode ultrasonography
Muscle architecture - fascicle length | Single time-point: 10 minutes
  Analysis of vastus lateralis fascicle length using b-mode ultrasonography

CONTACTS AND LOCATIONS:
Locations (1):
- Centre of Metabolism, Ageing and Physiology (COMAP), University of Nottingham, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No